CLINICAL TRIAL: NCT00479479
Title: Cobalamin Supplementation During Infancy; Effect on B-vitamin Status, Growth and Psychomotor Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); Foundation to Promote Research into Functional Vitamin B12 Deficiency, Bergen, Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16941
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Vitamin B 12 Deficiency
Keywords: cobalamin; methylmalonic acid; homocysteine; folate; newborns; infants; Deficiency Disease; Breastfeeding; Infant
MeSH Terms: conditions — Vitamin B 12 Deficiency; Deficiency Diseases; Breast Feeding | interventions — Hydroxocobalamin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cobalamin (Experimental): An intramuscular injection of 400 µg hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma, Norway)
  Interventions: Drug: Hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma)
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma) — an intramuscular injection of 400 µg hydroxycobalamin (Vitamin B12 Depot, Nycomed Pharma, Norway)
  Arms: Cobalamin

SUMMARY:
Adequate levels of vitamin B12 (cobalamin) is necessary for normal growth and development in infants. We have earlier investigated cobalamin status in healthy children and we observed metabolic evidence of impaired cobalamin status during the first 6 months, but not later in life.

The purpose of this study is to determine if cobalamin supplementation may influence the metabolic profile related to cobalamin status in infants.

DETAILED DESCRIPTION:
During fetal life and infancy, an adequate cobalamin status is important for normal growth and central nervous system development. A metabolic profile consistent with impaired cobalamin status is prevalent in breast-fed infants. Whether this profile reflects immature organ systems or cobalamin deficiency has not been clarified.

Low levels of cobalamin, elevated levels of total homocysteine (tHcy), cystathionine and/or methylmalonic acid (MMA) in the blood are measures of impaired cobalamin status.

The purpose of this randomized, controlled study is to determine if cobalamin supplementation may influence the metabolic profile related to cobalamin status in infants.

Six weeks old infants will be randomly assigned to receive either an intramuscular injection with 400 µg cobalamin or no intervention. Concentrations of cobalamin and folate in serum, and total homocysteine (tHcy), methylmalonic acid (MMA) and cystathionine in plasma will be determined at inclusion and at the age of 4 months. A questionnaire on infant and maternal nutrition, vitamin supplementation, growth parameters, parity and maternal use of tobacco will be completed.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks old infants
* The infant should be healthy and not have any serious malformations
* The mother should be healthy and not have any serious disorders or use any daily medications
* The mother should have an ordinary omnivorous diet

Exclusion Criteria:

* If there are evidence of serious infant disease during the study period, the infant should be excluded from the study

Ages: 4 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2004-12; Primary Completion 2006-08 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Measure: Outcome is related to changes in Cobalamin status: serum levels of cobalamin and folate, and the metabolic markers, plasma-tHcy, cystathionine and MMA | Infant age 6 weeks - 4 months

SECONDARY OUTCOMES:
Outcome is related to changes in growth parameters; weight, length, head circumference | Infant age: 6 weeks - 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Bjørke Monsen, M.D., Ph.D., Principal Investigator — Haukeland University Hospital
Locations (1):
- Laboratory of Clinical Biochemistry and Department of Pediatrics; Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Bjorke Monsen AL, Ueland PM, Vollset SE, Guttormsen AB, Markestad T, Solheim E, Refsum H. Determinants of cobalamin status in newborns. Pediatrics. 2001 Sep;108(3):624-30. doi: 10.1542/peds.108.3.624. PMID 11533328
- [Background] Monsen AL, Refsum H, Markestad T, Ueland PM. Cobalamin status and its biochemical markers methylmalonic acid and homocysteine in different age groups from 4 days to 19 years. Clin Chem. 2003 Dec;49(12):2067-75. doi: 10.1373/clinchem.2003.019869. PMID 14633879
- [Background] Allen LH. Vitamin B12 metabolism and status during pregnancy, lactation and infancy. Adv Exp Med Biol. 1994;352:173-86. doi: 10.1007/978-1-4899-2575-6_14. PMID 7832046
- [Background] Rosenblatt DS, Whitehead VM. Cobalamin and folate deficiency: acquired and hereditary disorders in children. Semin Hematol. 1999 Jan;36(1):19-34. PMID 9930566
- [Derived] Bjorke-Monsen AL, Torsvik I, Saetran H, Markestad T, Ueland PM. Common metabolic profile in infants indicating impaired cobalamin status responds to cobalamin supplementation. Pediatrics. 2008 Jul;122(1):83-91. doi: 10.1542/peds.2007-2716. PMID 18595990